CLINICAL TRIAL: NCT02287701
Title: Exploratory Investigation of Advanced PET/MRI Metrics for Bladder Cancer Characterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Society of Abdominal Radiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-00072
Record Dates: First submitted 2014-10-15; First posted 2014-11-11 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; MRI; PET
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MRI (Experimental): Patient receives MRI
  Interventions: Procedure: PET/MRI

INTERVENTIONS:
Procedure: PET/MRI — Simultaneous PET/MRI (3T system)
  Other Names: Siemens Biograph mMR

SUMMARY:
The overarching goal of this project is to explore whether associations exist between metrics obtained from PET/MRI incorporating advanced MRI sequences and features of bladder cancer, including grade, stage, and treatment response.

DETAILED DESCRIPTION:
The investigators will assess an advanced non-Gaussian diffusion-weighted imaging (DWI) model termed diffusion kurtosis imaging, multi-echo T2 mapping, dynamic contrast-enhanced (DCE) MRI using a motion-robust high-temporal and high-resolution radial acquisition scheme employing compressed sensing, and simultaneously acquired 18-fluoro (18F)- fluorodeoxygluclose (FDG) data. Preliminary data demonstrates the investigators ability to execute and evaluate all of these techniques at the investigators center. The investigators hypothesize that these techniques will be sensitive to functional and metabolic differences between subsets of bladder cancer cases and will improve upon the performance of current imaging protocols in bladder cancer characterization. Moreover, the investigators believe that these techniques will provide complementary information, such that they may be combined in a synergistic fashion for bladder cancer evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or imaging evidence of urothelial carcinoma of the bladder
* Age ≥ 18 years of age
* If female of childbearing potential, pregnancy test is negative. (In these instances, the patient will need to provide documentation of negative pregnancy test results.)

Exclusion Criteria:

* Inability to tolerate MRI including conditions such as claustrophobia or inability to lay flat for > 45 minutes.
* Presence of pacemaker/implantable cardiac device (ICD) or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Tumor standardized uptake value (SUV) from 18-fluorodeoxyglucose PET/MRI scan | within one week of study completion
  The tumor SUV value obtained approximately one hour following 18-fluorodeoxyglucose administration will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenkrantz, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States